CLINICAL TRIAL: NCT07385209
Title: Design and Application of a Home Care Mini-Program for Children With Congenital Heart Disease After Discharge: A Randomized Controlled Trial
Brief Title: Design and Application of a Home Care WeChat Mini-Program for Children After Congenital Heart Disease Surgery
Acronym: CHD-HomeCare
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ruijie YangLan (Other)
Responsible Party: Sponsor-Investigator, ruijie YangLan, Graduate Student, First Affiliated Hospital of Kunming Medical University
Organization: First Affiliated Hospital of Kunming Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025L393; 72364022 (Other: National Natural Science Foundation of China)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease
Keywords: home care; mobile health; postoperative rehabilitation; caregiver support
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the behavioral intervention (use of a specific WeChat mini-program), it was not feasible to blind the participants, care providers, or investigators. However, the outcomes assessors and data analysts were blinded to group allocation throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants receiving the WeChat mini-program intervention.
  Interventions: Other: Routine Care with Telephone Follow-up
- Control Group (Active Comparator): Participants receiving routine care with telephone follow-up.
  Interventions: Device: Home Care WeChat Mini-Program

INTERVENTIONS:
Device: Home Care WeChat Mini-Program — A family-centered WeChat mini-program providing health education, peer support, and remote monitoring for post-operative care.
  Arms: Control Group
Other: Routine Care with Telephone Follow-up — Participants in this group will receive standard post-discharge care as per hospital protocol, which includes initial discharge education and scheduled telephone follow-ups by hospital staff at 1, 3, and 6 months post-discharge to assess the child's status and answer questions.
  Arms: Intervention Group

SUMMARY:
This is a single-blind, randomized controlled trial aimed at evaluating the effectiveness of a family-centered, WeChat-based home care mini-program for children after congenital heart disease (CHD) surgery. Given the chronic nature of post-operative CHD management and the significant stress placed on families, this study shifts from a deficit-based to a strengths-based perspective, guided by the Double ABC-X model. Children (≤12 years old) who have undergone CHD surgery and their primary caregivers will be recruited. Participants will be randomly assigned to either the intervention group, which uses the mini-program for health education, peer support, and physiological monitoring, or the control group, which receives routine telephone follow-up. The primary outcomes are family health (measured by the Family Health Scale), family stress, and the quality of life for both the child and caregivers. Secondary outcomes include physiological parameters such as the 6-minute walk test distance. The study aims to provide evidence for a scalable digital health intervention to support long-term family adaptation and child recovery.

DETAILED DESCRIPTION:
1. Background and Rationale Congenital heart disease (CHD) is the most common birth defect globally, with a high prevalence in China. While surgical advances have significantly improved survival rates, CHD has transitioned into a chronic condition requiring long-term management. The post-discharge period places immense stress on families, affecting caregiver well-being, family functioning, and the child's recovery. Existing home care models often focus on the child's deficits or rely on resource-intensive methods (e.g., home visits). Guided by the Double ABC-X model of family adaptation, this study adopts a family strengths-based perspective. It aims to develop and test a digital, interactive home care mini-program designed to support family resources, promote positive adaptation, and improve health outcomes after CHD surgery.
2. Study Objectives Primary Objective: To evaluate the effectiveness of a family-centered, WeChat-based home care mini-program on improving family health in households with children after CHD surgery.

   Secondary Objectives: To assess the program's impact on: 1) reducing family stress, 2) enhancing the quality of life of both the child and primary caregivers, and 3) improving the child's physiological recovery indicators.
3. Study Design This is a prospective, two-arm, parallel-group, assessor-blinded, randomized controlled trial (RCT). Participants will be randomly assigned in a 1:1 ratio to either the intervention group or the control group.
4. Participants, Setting, and Timeline Participants: Families (the child who underwent surgery and their primary caregiver/parent) of children (≤12 years old) with CHD after surgical intervention.

   Setting: Recruitment and baseline assessment will be conducted at a tertiary hospital in Yunnan Province, China. The intervention and follow-up will be home-based.

   Sample Size: 210 families (105 per group), calculated with 80% power, a significance level of 0.05, an effect size (δ/σ) of 0.5, and accounting for 20% attrition.

   Timeline:

   Study Start Date (first enrollment): December 2025.

   Primary Completion Date (last participant's final data collection for primary outcome): December 2026.

   Study Completion Date: January 2027.
5. Interventions

   Intervention Group: Will receive access to the "CHD Postoperative Home Care" WeChat mini-program in addition to routine care. The mini-program includes three core modules:

   Education Module: Provides multimedia (text, images, video) health information on post-operative care, nutrition, medication, activity guidance, and complication monitoring.

   Interactive Support Module: Features a secure peer-support community for sharing experiences (digital narrative therapy) and a direct communication channel for families to consult the healthcare team.

   Monitoring & Alert Module: Allows families to log and submit key health data (e.g., weight, symptoms). The system includes automated alerts for concerning values and prompts for scheduled follow-up assessments. The research team will remotely monitor this data and initiate follow-up calls if alerts are triggered.

   Control Group: Will receive routine postoperative care, which includes standard discharge instructions and scheduled telephone follow-ups by hospital staff at 1, 3, and 6 months post-discharge.
6. Outcome Measures and Assessment Timepoints Assessments will occur at baseline (T0, pre-discharge) and at 1 (T1), 3 (T2), and 6 (T3) months post-discharge.

   Primary Outcomes:

   Family Health: Measured by the Chinese version of the Family Health Scale (FHS).

   Family Stress: Measured by the Congenital Heart Disease Family Stressor Scale.

   Quality of Life of Caregivers: Measured by the 36-Item Short Form Health Survey (SF-36).

   Quality of Life of the Child: Measured by the Chinese version of the Pediatric Quality of Life Inventory (PedsQL) Cardiac Module.

   Secondary Outcomes (Child Physiological Measures):

   Functional Capacity: 6-Minute Walk Test distance.

   Growth: Body weight.

   Cardiac Function: Heart rate and Left Ventricular Ejection Fraction (via echocardiogram).
7. Randomization, Blinding, and Data Analysis

   Randomization: After baseline assessment, eligible families will be randomly assigned using computer-generated random numbers sealed in opaque envelopes.

   Blinding: Outcome assessors and data analysts will be blinded to group allocation. Due to the nature of the intervention, participants and intervention facilitators cannot be blinded.

   Statistical Analysis: Data will be analyzed using SPSS software. Baseline characteristics will be compared using t-tests, chi-square, or Mann-Whitney U tests. Primary and secondary outcomes will be analyzed using Linear Mixed Models (LMM) for repeated measures to examine group, time, and interaction effects.
8. Ethical Considerations The study protocol has been submitted for approval to the Institutional Review Board of Kunming Medical University. Written informed consent will be obtained from all participating caregivers. The study will adhere to principles of confidentiality, beneficence, and the right to withdraw without penalty.

ELIGIBILITY:
Inclusion Criteria:

* - The child is ≤12 years old.
* The child has been diagnosed with congenital heart disease (CHD) and is scheduled for or has undergone corrective surgery.
* The child is in a stable medical condition (non-acute phase).
* At least one primary caregiver (parent or sibling >12 years old) of the child agrees to participate.
* The caregiver provides written informed consent to participate in the study.

Exclusion Criteria:

* - The child has severe developmental defects.
* The child has other major diseases that significantly affect quality of life.
* The caregiver has visual, hearing, or cognitive impairments that hinder communication.
* The caregiver has a diagnosed psychiatric disorder.
* The caregiver is unconscious or otherwise unable to provide consent.

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Family Health Score | Change from Baseline at 6 months post-discharge
  Score on the Chinese version of the Family Health Scale (FHS).
Family Stress Score | Change from Baseline at 6 months post-discharge
  Score on the Congenital Heart Disease Family Stressor Scale.
Child's Quality of Life Score | Change from Baseline at 6 months post-discharge
  Score on the Chinese version of the Pediatric Quality of Life Inventory (PedsQL) Cardiac Module.
Caregiver's Quality of Life Score | Change from Baseline at 6 months post-discharge
  Score on the 36-Item Short Form Health Survey (SF-36).

SECONDARY OUTCOMES:
Body Weight | Measured at 1, 3, and 6 months post-discharge
  Body weight measured in kilograms.
Left Ventricular Ejection Fraction | Measured at 6 months post-discharge
  Percentage measured by echocardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Ma,, professor of nursing, Principal Investigator — First Affiliated Hospital of Kunming Medical University; Fang Ma, professor of nursing, Principal Investigator — First Affiliated Hospital of Kunming Medical University
Locations (1):
- First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of pediatric and family health data, individual participant data will not be shared publicly to protect participant confidentiality.